CLINICAL TRIAL: NCT02566707
Title: Pharmacokinetics, Safety and Efficacy of Atazanavir /Dolutegravir/Lamivudine Regimen as Maintenance Regimen in Patients With Intolerance and/or Resistance to NRTIs, NNRTIs and RTV: A Pilot Study
Brief Title: Pharmacokinetics of Atazanavir /Dolutegravir/Lamivudine Regimen as Maintenance Regimen
Acronym: PRADAII
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to introduction of another integrase inhibitor, recruitement was not feasible anymore.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 14.08
Record Dates: First submitted 2015-09-02; First posted 2015-10-02 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Atazanavir Sulfate; dolutegravir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRADAII regimen (Experimental): Use of PRADAII regimen during 12 weeks. This regimen consists of atazanavir 400 mg QD, dolutegravir 50 mg QD, lamivudine 300 mg QD.
  Interventions: Drug: Atazanavir; Drug: Dolutegravir; Drug: Lamivudine

INTERVENTIONS:
Drug: Atazanavir — HIV therapy will be adapted: atazanavir 400mg QD
  Other Names: Reyataz
Drug: Dolutegravir — HIV therapy will be adapted: dolutegravir 50mg QD
  Other Names: Tivicay
Drug: Lamivudine — HIV therapy will be adapted: lamivudine 300mg QD
  Other Names: Epivir

SUMMARY:
During the past years the treatment of HIV-1 infection has transformed towards chronic treatment. Patients are being treated with antiretroviral drugs for many years and become older. The risk of developing side-effects due to long term antiretroviral therapy is therefore more and more likely. New alternative once-daily maintenance regimes are needed for those who are extensively pre-treated and experience side-effects or toxicity on standard treatment combinations. A possible once-daily, fully active maintenance regimen is the combination of atazanavir (unboosted), dolutegravir and lamivudine (PRADAII regimen). This combination is expected to be a safe, once-daily maintenance regimen with a favorable side-effect profile. The combination suits patients with intolerance and/or resistance to NRTIs, NNRTIs and ritonavir, who have a suppressed viral load. However, for this new combination the pharmacokinetic profile is unknown and there are no data on short-term and long-term safety and efficacy. This study wille therefore asses the pharmacokinetics, safety and efficacy in a small number of HIV-1 infected patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected as documented by positive HIV antibody test and confirmed by Western Blot.
* Subject is in need for a switch in maintenance regimen due to adverse effects, toxicities, simplification and/or resistance.
* Subject is at least 18 years of age at the day of screening.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* HIV-1 RNA < 40 copies/mL for at least 6 months on antiretroviral therapy prior to inclusion.
* Subject has no documented resistance mutations to PIs, INSTIs or lamivudine.

Exclusion Criteria:

* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* Inability to understand the nature and extent of the trial and the procedures required.
* Pregnant female (as confirmed by an HCG test performed less than 3 weeks before the first dose) or breast-feeding female.
* Abnormal serum transaminases determined as levels being > 5 times upper limit of normal.
* Renal failure determined as an estimated Glomerular Filtration Rate (eGFR) < 50 ml/min (MDRD-based).
* Concomitant use of medications that interfere with atazanavir, dolutegravir or lamivudine pharmacokinetics: oxcarbazepine, phenytoin, phenobarbital, carbamazepine, St. John's wort, rifampicin, clarithromycin, H2 receptor antagonists, proton pump inhibitors, irinotecan, midazolam, triazolam, buprenorphine, aprepitant, modafinil, imatinib, co-trimoxazole, other antiretroviral drugs.
* Concomitant use of medications that are contraindicated for use with atazanavir, dolutegravir or lamivudine: alfuzosin, dofetilide, pimozide, quetiapine, quinidine, bepridil, simvastatin, atorvastatin, lovastatin, sildenafil (as for use in pulmonary arterial hypertension), cladribine.
* Active hepatobiliary or hepatic disease (including chronic hepatitis B or C infection).
* Alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of atazanavir, dolutegravir and lamivudine | week 2
  Pharmacokinetic parameters of atazanavir, dolutegravir and lamivudine

SECONDARY OUTCOMES:
efficacy (viral load) | week 2, 6 and 12
  efficacy (viral load) of the combination of atazanavir, dolutegravir and lamivudine
number of adverse events | week 2, 6 and 12
  number of adverse events of the combination of atazanavir, dolutegravir and lamivudine

CONTACTS AND LOCATIONS:
Locations (4):
- University of Bonn, Bonn, Germany
- Netherlands (3):
  - Rijstate, Arnhem
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - St. Elisabeth, Tilburg

REFERENCES:
- See also: Abstract page 36 — http://regist2.virology-education.com/Abstractbook/2016_6.pdf